CLINICAL TRIAL: NCT07371949
Title: APLIKASI CHRONO- NUTRITION : PENGARUH FIBER JELLY TERHADAP RESPON GLUKOSA DARAH, KEKENYANGAN POST PRANDIAL, DAN WEIGH LOSS PADA WANITA OVERWEIGHT"
Brief Title: CHRONO-NUTRITION APPLICATION: THE EFFECT OF FIBER JELLY ON POST PRANDIAL BLOOD GLUCOSE, SATIETY AND WEIGHT LOSS AMONG OVERWEIGHT WOMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Surabaya State University (Other)
Responsible Party: Principal Investigator, Noor Rohmah Mayasari, Assistant Professor, Surabaya State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: No.004/UN38.10/EC.KEPK/HK.01.0
Record Dates: First submitted 2026-01-02; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obese Adults
Keywords: overweight
MeSH Terms: conditions — Overweight | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Fibre jelly was formulated using basil seeds, psyllium husk, rosella water extract, and carrageenan. Fibre jelly contained approximately 7.89 g of fibre in each pouch (~100 g).
  Interventions: Combination Product: Fiber jelly
- Placebo (Placebo Comparator): the control jelly was formulated using water and carrageenan as a gelling agent. Both types of jelly contained the same amount of stevia and fructose as sweeteners.
  Interventions: Combination Product: Fiber jelly

INTERVENTIONS:
Combination Product: Fiber jelly — Fibre jelly was formulated using basil seeds, psyllium husk, rosella water extract, and carrageenan, while the control jelly was formulated using water and carrageenan as a gelling agent. Both types of jelly contained the same amount of stevia and fructose as sweeteners. Fibre jelly contained approximately 7.89 g of fibre in each pouch (~100 g).
  Other Names: Intervention

SUMMARY:
The goal of this observational study is to learn about the effects of pre meal fiber jelly in overweight women over the age of 20-60 who take intervention pre meal fiber jelly on their postprandial blood glucose level and appetite level.

The main question it aims to answer is:

Does pre meal fiber jelly in overweight women effect on their postprandial blood glucose level and appetite level?

DETAILED DESCRIPTION:
Prior to the test days, participants were asked to fast overnight following the standard procedure for fasting blood glucose measurement. Additionally, participants were asked to refrain from vigorous physical activity prior to the test days. On the test days, fasting blood glucose was taken prior to the breakfast test meal at 0 minute. Then, participants were asked to consume fibre jelly for those in the intervention group and carrageenan-based jelly for those in the control group. After consuming jelly, participants from both groups were asked to consume bread, which was equal to 50 grams of starch and 250 ml of water in 10 minutes. To measure their postprandial blood glucose levels, participants were required to fast for the next 2 hours. After blood samples were collected, participants were provided with a complete meal and unlimited water. Participants were allowed to eat and drink as much as they desire following their satiety and hunger cues (ad-libitum). The remaining foods were weighed to calculate the total calories consumed by participants.

ELIGIBILITY:
Inclusion Criteria:

(1) female adults aged between 20-60 years; (2) having fasting blood glucose level <125 mg/dL; (3) having body mass index (BMI) more than or equal to 23; (4) not undergoing loss weight program during the recruitment process; (5) not allergic to rosella and basil seed

Exclusion Criteria:

Candidates were excluded if they were pregnant or lactating, had any medical conditions, including gastrointestinal disorders, cardiovascular disease, or other chronic diseases, smoking, or consuming alcohol.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the study enrolls only biological females
Enrollment: 28 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-12-14 (Actual); Study Completion 2025-12-14 (Actual)

PRIMARY OUTCOMES:
Blood Glucose level | 0, 30, 45, 60, 90, 120 minute
  Post prandial blood glucose level
Appetite level | 0 minute, 30 minute, 45 minute, 60 minute, 90 minute, 120 minute, 180 minute, 240 minute
  Visual analog scale of hunger, fullness, appetite, prospective food, and satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports and Health Sciences, Surabaya, Indonesia, Indonesia

IPD SHARING:
Plan to Share IPD: No
The data will not shared to protect respondent privacy

DOCUMENTS (1):
  • Study Protocol (2026-01-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT07371949/Prot_000.pdf